CLINICAL TRIAL: NCT04636983
Title: A Phase I, Single-centre, Double-blind, Randomised, Placebo-controlled Clinical Trial to Investigate the Safety, Tolerability and Pharmacokinetics of BV100 Administered as Single Intravenous Doses to Healthy Male Subjects
Brief Title: Clinical Trial to Investigate the Safety, Tolerability and Pharmacokinetics of BV100 in Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: BioVersys SAS (Industry)
Responsible Party: Sponsor
Organization: BioVersys AG (Industry)
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BV100-01
Record Dates: First submitted 2020-11-10; First posted 2020-11-19 (Actual); Last update posted 2022-02-08 (Actual); Status verified 2021-10

CONDITIONS: Healthy Subjects

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BV100 (Experimental): BV100 intravenous infusion
  Interventions: Drug: BV100
- Placebo (Placebo Comparator): Saline intravenous infusion
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BV100 — Rifabutin IV
  Arms: BV100
Drug: Placebo — Saline
  Arms: Placebo

SUMMARY:
This is a Phase 1, single-centre, double-blind, randomised, placebo-controlled study to evaluate the safety, tolerability, and pharmacokinetics of single intravenous ascending doses of BV100 to healthy male subjects.

DETAILED DESCRIPTION:
The purpose of this First in human study is to evaluate the safety, tolerability, and pharmacokinetics of single intravenous ascending doses of BV100 to healthy subjects. Participants will either receive one single intravenous infusion of BV100 or placebo (physiological saline 0.9% w/v).

ELIGIBILITY:
Inclusion Criteria:

1. Subject must be 18 to 55 years of age inclusive at the time of signing the informed consent.
2. Subjects who are healthy as determined by the Investigator based on medical evaluation including medical history, physical and neurological examination, vital signs, ECG, and clinical laboratory tests at screening and on Day -1.
3. Subjects are able to have an intravenous line placed.
4. Body weight of at least 50 kg and BMI within the range of 19 to 30 kg/m2 (inclusive) at screening examination.
5. Male subjects will be included in the study.
6. Subjects must agree to the following from the time of the first dose until 3 months after the follow-up visit:

   * use two acceptable methods of birth control with a female partner of child-bearing potential (barrier method combined with an additional highly effective contraceptive method). Barrier methods of contraception include condom or occlusive cap (diaphragm or cervical/vault caps). Highly effective contraception is defined in accordance with the Clinical Trial Facilitation Group (CTFG 2014 ) guidance and includes the following methods: implants, injectables, hormonal intrauterine device, combined hormonal contraceptives, sexual abstinence and vasectomized sexual partner.
   * refrain from donating sperm.
7. Prior to any clinical study specific procedure the subject provided written informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol. Subjects must be able to read, write, and fully understand the German language.

7. Prior to any clinical study specific procedure the subject provided written informed consent as described in Appendix 3 which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol. Subjects must be able to read, write, and fully understand the German language.

Exclusion Criteria:

1. History of clinically relevant disease of any organ system that may interfere with the objectives of the study or provide a risk to the health of the subject.
2. Known or suspected history of hypersensitivity to rifabutin or excipients or to drugs of a similar chemical class including rifampicin, rifapentine, rifaximin; history of allergic reactions leading to hospitalisation or any other allergic conditions (including drug allergies, asthma, eczema, anaphylactic reactions but excluding untreated, asymptomatic, seasonal allergies) which the Investigator considers may affect the safety of the subject and/or outcome of the study.
3. History of antibiotic associated diarrhoea within the last year.
4. History of epilepsy, other neurological disorders, or neuropsychiatric conditions.
5. Subjects with ECG abnormalities (history, or evidence of second-degree heart block of Mobitz type II, third degree heart block, or any abnormality considered relevant by the Investigator), QTcF > 450 ms, PR > 200 ms, or QRS duration > 110 ms.
6. Supine systolic blood pressure > 140 mmHg or < 90 mmHg or diastolic blood pressure > 90 mmHg or < 50 mmHg at Screening or Day 1 prior to dosing (any abnormal blood pressure results may be repeated once and if the repeat result is within the normal range, it is not considered to have met the exclusion criterion). Pulse rate > 90 or < 50 beats per minute at Screening or Day 1 prior to dosing.
7. Glomerular Filtration Rate (GFR) < 90 mL/min/1.73m2 as calculated by the Chronic Kidney Disease Epidemiology Collaboration formula. In case of a borderline result between ≥ 80 and < 90 mL/min, Cystatin C will be determined in addition, and the subject will only be included if the Cystatin C value is below the upper limit of normal (ULN).
8. Alanine aminotransferase (ALT), aspartate aminotransferase (AST), alkaline phosphatase (ALP) and creatinine, above the ULN at Screening. Any abnormal value of these parameters may be repeated and if the repeat result is within the laboratory reference range, it is not considered to have met the exclusion criterion.
9. Screening values other than AST, ALT, ALP, creatinine, for haematology, biochemistry, or urinalysis must not exceed the reference range. Minor deviations from normal are allowed, if they are not clinically significant.
10. History of symptomatic, chronic or recurrent infection (e.g. nausea, vomiting, diarrhoea, infection with fever) or any viral (including symptomatic herpes zoster), bacterial (including upper respiratory infection), fungal (non-cutaneous) or parasitic infection within 30 days prior to admission to the clinical unit.
11. Subjects who have received any prescribed systemic or topical medication within 4 weeks of the dose administration or within 5 times the half-life, whichever is longer, except for the occasional use of paracetamol (up to 2 g/day).
12. Subjects who have used any non-prescribed systemic or topical medication (including dietary supplements, natural and herbal remedies) or megadose vitamins (i.e. 20 to 600 times the recommended daily supplement dose) within 7 days of the dose administration, unless in the opinion of the Investigator the medication will not interfere with the study procedures or compromise safety.
13. Subjects who have received any medications, including St John's Wort, known to chronically alter drug absorption or elimination processes within 30 days of the first dose administration.
14. Regular use of any inducer of metabolism (e.g., barbiturates, rifampin) in the 3 months prior to the first admission to the clinical unit.
15. Administration of live vaccine(s) within 1 month prior to screening, or plans to receive such vaccines during the study.
16. Subjects who have participated in a clinical study involving administration of an investigational drug (new chemical entity) within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
17. Exposure to more than 4 new chemical entities in the last 12 months before the first dosing day in this study.
18. A positive pre-study serology test for hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibodies or human immunodeficiency virus (HIV)-1 and/or 2 antibodies.
19. A positive pre-study drug/alcohol screen.
20. Subjects who consume more than 21 units of alcohol per week or who have a significant history of alcoholism or drug/chemical abuse (one unit of alcohol equals ½ pint [285 mL] of beer or lager, one glass [125 mL] of wine, or 30 mL of 40% of alcohol by volume distilled spirits).
21. Excessive consumption of caffeine- or xanthine-containing food or beverages (> 5 cups of coffee a day or equivalent) or inability to stop consuming from 48 hours prior to study treatment administration.
22. Any use of drugs-of-abuse or alcohol abuse within 2 years prior to the first admission to the clinical unit.
23. Subjects who are unable to refrain from the consumption of Seville oranges, grapefruit or grapefruit juice and /or pomelos, exotic citrus fruits, grapefruit hybrids, starfruit or fruit juices from 1 day prior to the first dose of Study Drug on Day 1, until completion of the last PK blood sample time point.
24. Inability to understand or communicate reliably with the Investigator or considered by the Investigator to be unable to or unlikely to co-operate with the requirements of the study.
25. Any other conditions or factors which in the opinion of the Investigator may interfere with study conduct. Failure to satisfy the Investigator of fitness to participate for any other reason.
26. Any significant blood loss, donated one unit (450 mL) of blood or more, or received a transfusion of any blood or blood products within 60 days, or donated plasma within 7 days prior to the first admission to the clinical unit.
27. Inability to refrain from using soft contact lenses starting from administration of study treatment until follow-up visit.
28. Subjects who are study site employees or immediate family members of the study site or Sponsor employee.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — • Healthy male subjects
Enrollment: 54 (Actual)
Dates: Start 2020-11-09 (Actual); Primary Completion 2021-12-12 (Actual); Study Completion 2022-01-20 (Actual)

PRIMARY OUTCOMES:
To investigate the safety and tolerability of single intravenous ascending doses of BV100 assessed by the nature, occurrence, and severity of treatment-emergent adverse events | 10 Days
  Safety and tolerability

SECONDARY OUTCOMES:
To characterize the single dose pharmacokinetic profile of rifabutin: Area under the plasma concentration versus time curve (AUC) | 120 hours
  Pharmacokinetics
To characterize the single dose pharmacokinetic profile of rifabutin: Peak Plasma Concentration (Cmax) | 120 hours
  Pharmacokinetics

OTHER OUTCOMES:
To determine the urinary excretion of BV100: Cumulative amount excreted within 24 and 96 hours after start of infusion | 96 hours
  Pharmacokinetics
To determine the plasma concentration of the main metabolite 25-O-Desacetyl-Rifabutin in plasma | 5 days
  Pharmacokinetics

CONTACTS AND LOCATIONS:
Overall Officials: Denis Strugala, MD, Principal Investigator — Nuvisan GmbH
Locations (1):
- Nuvisan GmbH, Neu-Ulm, Germany

IPD SHARING:
Plan to Share IPD: No